CLINICAL TRIAL: NCT06085391
Title: Testing the Efficacy of the REThink Emotions Platform in a Full-scale SMART Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: REThink SMARTrial
Record Dates: First submitted 2023-10-06; First posted 2023-10-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REThink game (Experimental): Each recruited participant randomized in the experimental group will receive the REThink game app.
  Interventions: Other: REThink Game
- MoodWheel (Active Comparator): The participants randomized in the control group will complete the MoodWheel app.
  Interventions: Other: MoodWheel
- PsyPills (Experimental): Participants from experimental group who do not respond to REThink game alone will receive the PsyPills app
  Interventions: Other: REThink Game; Other: PsyPills

INTERVENTIONS:
Other: REThink Game — REThink Game is the therapeutic game that uses psychological science to help youths find their superhero emotional strengths! It is composed of seven levels, each training a specific emotion regulation ability: emotion recognition, mindfulness and relaxation, cognitive change, positive bias, distinction between useful and useless thoughts, problem solving and compassion.
  Arms: PsyPills; REThink game
Other: MoodWheel — Mood Wheel is a web and mobile-based app that uses experience sampling procedures for the assessment of current/previous distress and positive emotions. The aim of the app is to inquire about the valence, control and functionality of users' emotions.
  Arms: MoodWheel
Other: PsyPills — PsyPills is a self-help psycho-educational instrument intended to build stress resilience and to target (only) mild and transient negative mood states, alone or in combination with other methods/instruments.
  Psychological Pills (PsyPills) are inspired by Rational-Emotive & Cognitive-Behavioral Therapy (CBT/REBT), which has strong evidence for its efficacy/effectiveness in human development/health promotion and in the treatment of a variety of psychological conditions.
  The PsyPills app was tested in a pilot study and showed positive effects on reducing distress.
  Arms: PsyPills

SUMMARY:
This activity will have the objective of testing the validity of the integrated in-game assessment and personalized REThinkEMOTIONS platform in the prevention of emotional disorders in youth.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents between 8 and 16 years old
* provided written parental consent
* able to access mobile/internet applications on their device

Exclusion Criteria:

* Intellectual disability or physical limitations precluded the use of the computer program
* Had a major mental health disorder

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Levels of rational and irrational beliefs | baseline, pre-intervention
  The Child and Adolescent Scale of Irrationality will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Changes of rational and irrational beliefs | Post-intervention (one week after the intervention)
  The Child and Adolescent Scale of Irrationality will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Fluctuations in of rational and irrational beliefs | 6 months Follow-up
  The Child and Adolescent Scale of Irrationality will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Levels of emotion-regulation | baseline, pre-intervention
  The Emotion Regulation Index for Children and Adolescents (ERICA) It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Changes in emotion-regulation | Post-intervention (one week after the intervention)
  The Emotion Regulation Index for Children and Adolescents (ERICA). It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Fluctuations in emotion-regulation | 6 months Follow-up
  The Emotion Regulation Index for Children and Adolescents (ERICA). It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Levels of child behavioral difficulties | Pre-intervention (one week before the intervention)
  Strengths and Difficulties Questionnaire (SDQ) is a self-report scale that measures emotional and behavioral difficulties in children and adolescents. Its is composed of items and 25 items ranked on a three points Liker scale from "not true" to "almost true". Greater scores at this scale represent higher level of difficulties.
Changes in child behavioral difficulties | Post-intervention (one week after the intervention)
  Strengths and Difficulties Questionnaire (SDQ) is a self-report scale that measures emotional and behavioral difficulties in children and adolescents. Its is composed of items and 25 items ranked on a three points Liker scale from "not true" to "almost true". Greater scores at this scale represent higher level of difficulties.
Fluctuations in child behavioral difficulties | 6 months follow-up
  Strengths and Difficulties Questionnaire (SDQ) is a self-report scale that measures emotional and behavioral difficulties in children and adolescents. Its is composed of items and 25 items ranked on a three points Liker scale from "not true" to "almost true". Greater scores at this scale represent higher level of difficulties.

SECONDARY OUTCOMES:
Level of emotional distress | baseline, pre-intervention
  The Profile of Emotional Distress (PED) is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Changes in emotional distress | Post-intervention (one week after the intervention)
  The Profile of Emotional Distress is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).
Fluctuations in emotional distress | 6 months follow-up
  The Profile of Emotional Distress is a is a 40-item self-report instrument measuring functional and dysfunctional negative emotions based on Albert Ellis's binary model of distress, as well as positive emotions. The negative emotion subscales include two dysfunctional emotion dimensions (anxiety and depression) and two functional counterparts (concern and sadness). Responders are asked to assess the degree to which they have experienced each emotion during the previous two weeks, based on a five-point Likert scale ranging from "Not at all" (0) to "Extremely" (4).

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No